CLINICAL TRIAL: NCT00520702
Title: A Randomized Trial to Compare Time to Common Toxicity Criteria for Adverse Effect (CTC AEC) 3.0 Grade. 3 Treatment Related Pneumonitis (TRP) in Patients With Locally Advanced Non-Small Cell Lung Carcinoma (NSCLC) Receiving Concurrent Chemoradiation Radiation Treated With 3-Dimensional Conformal Radiation Therapy (3D CRT, ARM 1) Versus Intensity Modulated Radiation Therapy (IMRT, ARM 2) Using 4-Dimensional CT Planning and Image Guided Adaptive Radiation Therapy (IGART)
Brief Title: 3-Dimensional Conformal Radiation Therapy Versus Intensity Modulated Radiation Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2006-0222; NCI-2012-01595 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-08-22; First posted 2007-08-24 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Lung Cancer; 3-Dimensional Conformal Radiation Therapy; Intensity Modulated Radiation Therapy; 3D CRT; IMRT; NSCLC; TRP; Treatment related pneumonitis
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy, Intensity-Modulated; Radiotherapy, Conformal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 3D CRT (Active Comparator): 3-Dimensional Conformal Radiation Therapy (3D CRT)
  Interventions: Procedure: 3-Dimensional Conformal Radiation Therapy
- IMRT (Active Comparator): Intensity-Modulated Radiation Therapy (IMRT)
  Interventions: Procedure: Intensity Modulated Radiation Therapy

INTERVENTIONS:
Procedure: Intensity Modulated Radiation Therapy — 66 Gy in 33 Daily Fractions at 2 Gy per fraction.
  Other Names: IMRT
  Arms: IMRT
Procedure: 3-Dimensional Conformal Radiation Therapy — 66 Gy in 33 Daily Fractions at 2 Gy per fraction.
  Other Names: 3D CRT
  Arms: 3D CRT

SUMMARY:
Primary Objective:

* Developing Common Toxicity Criteria (CTC) 3.0 grade > 3 treatment related pneumonitis (TRP) or
* Developing local-regional recurrence among patients treated with 3D conformal radiation therapy (CRT) (Arm 1) or intensity modulated radiation therapy (IMRT) (Arm 2).

Secondary Objectives:

* To assess and compare the time to develop CTC 3.0 grade > 3 radiation esophagitis in patients with non-small cell lung cancer (NSCLC) treated in arm 1 and arm 2.
* To investigate the association of inflammatory cytokines with the time to the development of radiation pneumonitis and outcomes to concurrent chemoradiation between arm 1 and arm 2.
* To investigate the association of relevant pharmacogenetics, biomarkers, and gene polymorphisms with the time to the development of radiation pneumonitis and treatment outcomes to concurrent chemoradiation between arm 1 and arm 2.
* To evaluate image guided adaptive radiation therapy (IGART) using weekly computed tomography (CT) on rail or cone beam CT in the assessment of tumor response and impact on treatment planning and delivery.
* To compare overall survival, progression-free survival, median survival time, in arm 1 and arm 2.
* To evaluate the role of functional image of fluorodeoxyglucose-positron emission tomography (FDG-PET) in assessing and predicting the time to the development of TRP and tumor response.
* To measure and compare symptom burden over time of the treatment using MD Anderson Symptom Inventory (MDASI)-Lung in the 2 arms.
* To determine the impact of comorbid conditions on survival.

DETAILED DESCRIPTION:
TRP (treatment related pneumonitis) is an inflammation (irritated or injured tissue) of the lungs that occurs as a result of chemotherapy or radiation therapy. TRP occurs because both chemotherapy and radiation affect normal lung tissue when tumors are being treated.

3D CRT is the current standard of care. It delivers radiation to several different angles of the body with center focus on the tumor(s). Because it is delivered at different angles, the same amount of radiation that contacts the tumor(s) also contacts normal lung tissue at each angle.

IMRT is a new type of radiation therapy. It also delivers radiation to several different angles of the body with center focus on the tumor(s). The difference is that the amount of treatment at each angle is adjusted according to the shape and size of the tumor(s), which in turn may decrease radiation exposure to normal lung tissue at each angle. Researchers want to find out if intensity modulated radiation therapy (IMRT) is able to decrease the amount of normal lung that is affected when treating lung cancer.

Before you can start treatment on this study, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. You will have a physical exam, including measurement of your vital signs (blood pressure, heart rate, temperature, and breathing rate). You will have blood drawn (about 1 tablespoon) and urine collected for routine tests. You will be asked about any other medical problems you may have that could cause the development of TRP. You will have tests that include a computed tomography (CT) scan, positron emission tomography (PET) scan, and lung function test. A PET scan is a scan that will show cells that take in higher levels of a type of sugar (glucose), such as cancer cells. Before the scan, a small dose of a slightly radioactive form of glucose will be injected through a vein. The cells that take in higher amounts of glucose will show up better on the scan. The scanning process is quite similar to a regular CT scan. No new biopsy is needed; only the original biopsy will be used for this study.

You will have 2 different single photon-emission computed tomography tests (SPECTs). You will have a lung single-photon emission computerized tomography (SPECT)test that will show the area of blood flow in the normal lung. You will have a heart single-photon emission computerized tomography (SPECT) test that will show the areas of blood flow in the heart. To perform these single-photon emission computerized tomography (SPECT) tests, you will have a slightly radioactive substance injected into your vein so that images can be seen of the blood flow in the lung and heart. This will help the study doctor try to avoid using radiation angles that would go through the normal blood flow area. You will also have a biopsy of your tumor tissue. To perform a tumor biopsy, an area of the body (where tumor is present) is numbed with anesthetic, and a small amount of tumor tissue is withdrawn through a large needle or with forceps (a tong-like instrument) during an endoscopic (viewing of body cavity with a special instrument) exam.

Researchers will use the results of these tests to learn the stage (size and location) of the cancer to see if the tumor(s) can be treated by radiation. Women who are able to have children must have a blood or urine pregnancy test, which will be performed on the same blood or urine that was collected for routine tests. To be eligible to take part in this study, the pregnancy test must be negative.

If you are found to be eligible to take part in this study, your radiation doctor will first conduct a planning session. You will have a CT scan of your chest, and your respiratory (breathing) motion will be monitored. After the scan is done, your radiation doctor will evaluate it and make an outline of the tumor(s) in your lung. The CT scan helps the doctor identify (note the difference between) the tumor(s) and the normal surrounding tissue. The planning session helps the radiation doctor decide the target area(s), the best angles to deliver the radiation, and the most effective radiation dose (which is also intended to decrease radiation to surrounding normal tissues) for treatment.

If the plan for treatment is considered acceptable for you by the radiation doctor, you will then be randomly assigned (as in the toss of a coin) to 1 of 2 treatment groups. Participants in one group will receive 3D CRT. Participants in the other group will receive intensity modulated radiation therapy (IMRT). You will have an equal chance of being in either one of these groups. If you are assigned to receive intensity modulated radiation therapy (IMRT), the total radiation dose to the tumor(s) will be slightly higher than for participants receiving 3D CRT.

If the 3D CRT plan for treatment is not considered acceptable for you (usually because of a large target area) by the radiation doctor, you will be treated with IMRT, with or without amifostine. Amifostine is a drug given as an injection to protect the normal lung and esophagus tissue from radiation side effects and injury. Your treating physician will decide if you need amifostine or not, based on the size of the tumor tissue and normal tissue in the radiation "field" (the area given radiation during treatment). If you need amifostine, a nurse will give you the injection about 30 minutes before radiation treatment. Your blood pressure will be checked for 15-20 minutes after injection.

Participants on this study will be receiving standard chemotherapy given together with radiation therapy. The standard chemotherapy usually includes cisplatin, carboplatin, paclitaxel, or docetaxel. The chemotherapy is not considered the investigational part of this study.

All study participants will receive standard chemotherapy, given together with radiation therapy. The standard chemotherapy usually includes cisplatin, carboplatin, paclitaxel, and/or docetaxel. Your chemotherapy doctor will explain the side effects of these chemotherapy drugs to you before you start receiving chemotherapy. The chemotherapy is not the investigational part of this clinical trial.

Participants in each group will receive a total of 6 ½ weeks of radiation therapy (once a day for 5 days a week). You will not be treated on the weekends or on a national holiday. If the disease gets worse or you experience any intolerable side effects, you will be taken off this study.

After you have completed therapy on this study, you will have follow-up visits. The study doctor will check how the disease responded to treatment using the same imaging scans and blood tests (about 1 tablespoon each time) that were performed during the screening portion of this study. These tests will be performed about every 3-4 months after completion of treatment as part of your standard of care.

This is an investigational study. Both 3D conformal radiation therapy (CRT) and intensity modulated radiation therapy (IMRT) are FDA approved for the treatment of cancer. Up to 168 patients will take part in this study. All will be enrolled at M.D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically proven diagnosis of unresected loco-regionally advanced non-small cell lung cancer without evidence of hematogenous metastases, Stages IIB-IIIB without contralateral hilar nodal disease.
2. Patient is suitable for concurrent chemoradiation therapy per treating physician's assessment (kps >/= 70, weight loss < 10% in three months prior to diagnosis).
3. Patients with Stage IV NSCLC with solitary metastasis (brain, one side of adrenal gland, or one site of bone), who have clinical indication of concurrent chemoradiation to the primary disease in the lung are eligible.
4. Patients who received induction chemotherapy and then referred for concurrent chemoradiation are eligible.
5. Patients who had local regional recurrence after surgical resection and who are suitable for definitive concurrent chemoradiation are eligible.
6. Measurable disease by chest x-ray and/or contrast-enhanced CT, and/or PET scan
7. FEV 1> 1000 cc
8. Pre-chemoradiation FDG-PET within 10 weeks prior to randomization. This PET/CT is a standard procedure for staging. It is strongly encouraged to have this PET/CT performed at the same time for 4-D CT simulation using the 4-D PET/CT scanner at the department of radiation oncology.
9. Patient will undergo routine standard pretreatment evaluations as decided by treating physician, which usually include magnetic resonance imaging (MRI) or CT of the brain, contrast CT scan of the thorax and upper abdomen, pulmonary functional test, single-photon emission computerized tomography (SPECT), liver function tests (LFT), blood chemistry, renal functional test, complete blood count.
10. Age > 18, < 80 years
11. Patient must sign study specific informed consent prior to study entry.

Exclusion Criteria:

1. Evidence of small cell histology
2. Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
3. Pregnant women are ineligible as the treatment involves unforeseeable risks to the participant and to the embryo or fetus. Patients with childbearing potential must practice appropriate contraception.
4. Patient has enrolled in a clinical trial that specifically does not allow IMRT treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2007-08-21 (Actual); Primary Completion 2018-10-03 (Actual); Study Completion 2018-10-03 (Actual)

PRIMARY OUTCOMES:
Time to Treatment Failure | 3 months after radiation therapy
  Time to treatment failure defined as from the time of randomization to the development of treatment related pneumonitis (TRP) or local-regional recurrence, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Zhongxing Liao, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org